CLINICAL TRIAL: NCT05025566
Title: Cognitive Phenotyping of Severe Psychiatric Disorders
Brief Title: Cognitive Phenotyping of Severe Psychiatric Disorders (PSYCOG)
Acronym: PSYCOG
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: PSYCOG
Record Dates: First submitted 2021-07-19; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-07

CONDITIONS: Severe Psychiatric Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Psychotic disorders
  Interventions: Diagnostic Test: Cognitive (behavioural and neurophysiological) screening
- Depressive disorders
  Interventions: Diagnostic Test: Cognitive (behavioural and neurophysiological) screening
- Bipolar disorders
  Interventions: Diagnostic Test: Cognitive (behavioural and neurophysiological) screening
- Anxiety disorders
  Interventions: Diagnostic Test: Cognitive (behavioural and neurophysiological) screening
- Autism spectrum disorders
  Interventions: Diagnostic Test: Cognitive (behavioural and neurophysiological) screening
- Eating disorders
  Interventions: Diagnostic Test: Cognitive (behavioural and neurophysiological) screening
- Healthy volunteers
  Interventions: Diagnostic Test: Cognitive (behavioural and neurophysiological) screening

INTERVENTIONS:
Diagnostic Test: Cognitive (behavioural and neurophysiological) screening — Cognitive disorders are attested at the behavioral level by the psychologist specialized in neuropsychology who makes the patient take a standardized battery of specific psychometric tests. This assessment thus makes it possible to obtain behavioral data such as reaction time, error rates and modeling parameters.
  The electroencephalogram (EEG) consists of collecting the signal of the brain's bioelectrical activity by means of electrodes placed on the scalp. The EEG is used to determine the cerebral functioning underlying cognitive functions by performing it simultaneously with the behavioral tasks of the neuropsychological assessment, thus obtaining a neurophysiological phenotyping of cognitive disorders.

SUMMARY:
The identification of transnosographic dimensions constituted by cognitive disorders constitutes a particularly promising avenue for classifying psychiatric disorders in a more precise and personalized manner. However, despite interesting preliminary data, there is no exhaustive phenotyping of the different cognitive disorders in large samples where all severe psychiatric disorders are represented. Moreover, the brain mechanisms underlying cognitive disorders remain poorly understood, whereas their identification would allow a better understanding of the pathophysiology of these disorders as well as the identification of potential therapeutic targets.

Here, the investigators will compare cognitive-behavioral performance in patients with different types of severe psychiatric disorders (psychotic disorders, depressive disorders, bipolar disorder, anxiety disorders, autism spectrum disorders and eating disorders) and healthy volunteers to identify specific and shared cognitive alterations between the different severe psychiatric disorders. In addition, the investigators will compare neurophysiological cognitive data in to identify alterations in neurophysiological cognitive mechanisms that are specific to and shared between the different severe psychiatric disorders.

The investigators will include 180 patients suffering from a severe psychiatric disorder (psychotic disorder, mood disorder (depressive and bipolar disorders), anxiety disorder, autism spectrum disorder and eating disorder) and benefiting from cognitive phenotyping (neuropsychological assessment and possibly EEG) as part of the initial assessment for a severe psychiatric disorder. In parallel, the investigators will include 180 healthy volunteers The different variables corresponding to the judgment criteria will be compared between the groups by being included as dependent variables in mixed linear regression models (ANOVA; or KRUSKAL-WALLIS if non-parametric) with the group as independent factor, time (before, after treatment) and type of treatment.

This study will allow the constitution of a transnosographic atlas of neuro-cognitive deficits in different psychiatric pathologies.

DETAILED DESCRIPTION:
* Context : The identification of transnosographic dimensions constituted by cognitive disorders constitutes a particularly promising avenue for classifying psychiatric disorders in a more precise and personalized manner. However, despite interesting preliminary data, there is no exhaustive phenotyping of the different cognitive disorders in large samples where all severe psychiatric disorders are represented. Moreover, the brain mechanisms underlying cognitive disorders remain poorly understood, whereas their identification would allow a better understanding of the pathophysiology of these disorders as well as the identification of potential therapeutic targets.
* Method: Research involving the human being, prospective observational, monocentric (CHU Grenoble Alpes).
* Main objective : to compare cognitive-behavioral performance in patients with different types of severe psychiatric disorders (psychotic disorders, depressive disorders, bipolar disorder, anxiety disorders, autism spectrum disorders and eating disorders) and healthy volunteers to identify specific and shared cognitive alterations between the different severe psychiatric disorders. The primary outcome is the comparison of cognitive-behavioral performance composite scores corresponding to response rates (in %) for each cognitive dimension between the different severe psychiatric disorder groups and the healthy subjects.
* Secondary objective 1: The first secondary objective of PSYCOG is to compare neurophysiological cognitive data in patients with different types of severe psychiatric disorders (psychotic disorders, depressive disorders, bipolar disorder, anxiety disorders, autism spectrum disorders and eating disorders) and healthy volunteers to identify alterations in neurophysiological cognitive mechanisms that are specific to and shared between the different severe psychiatric disorders. Outcome will be the comparison of neurophysiological data from EEG recordings (evoked potentials, spectral dynamics, and brain source) recorded simultaneously with the performance of behavioral tasks for each cognitive dimension between the different severe psychiatric disorder groups and healthy subjects.
* Secondary objective 2: The second secondary objective of PSYCOG is to compare cognitive behavioral performance before and after treatments recommended and routinely prescribed to patients evaluated for a severe psychiatric disorder (psychotropic drug treatment, non-invasive neurostimulation, psychotherapy, psychoeducation, depending on the case) within the different groups of patients with severe psychiatric disorders. Outcome will be the comparison of behavioral data (response rates, reaction times, modeling parameters) from neuropsychological tests before and after treatment (up to + 6 months) in the different groups of patients with severe psychiatric disorders.
* Secondary objective 3: The third secondary objective of PSYCOG is to compare the neurophysiological cognitive data associated with cognitive behavioral tests before and after treatments recommended and routinely practiced in patients evaluated for a severe psychiatric disorder (psychotropic drug treatment, non-invasive neurostimulation, psychotherapy, psychoeducation as the case may be) within the different groups of patients with severe psychiatric disorder. Outcome will be the comparison of neurophysiological data obtained from EEG recordings (evoked potentials, spectral dynamics and brain source) associated with behavioral tests before and after treatment (up to + 6 months) in the different groups of patients with severe psychiatric disorder.
* Inclusion criteria for patients: 18 to 65 years of age, patients suffering from a severe psychiatric disorder (psychotic disorder, mood disorder (depressive and bipolar disorders), anxiety disorder, autism spectrum disorder and eating disorder), patient benefiting from cognitive phenotyping (neuropsychological assessment and possibly EEG) as part of the initial assessment for a severe psychiatric disorder, proven non-opposition to participation in the study, ability to perform cognitive tests: speaking and understanding French easily, presence of an identified support person, absence or presence of a property protection measure such as curatorship or guardianship
* Inclusion criteria for healthy volunteers: between the ages of 18 and 65, proven non-opposition to participating in the study, ability to perform cognitive tests: able to speak and understand French
* Non inclusion criteria: impossible to collect information on exposure (subjects recently arrived in France, foreign language ...), history of coma, epilepsy, head trauma with loss of consciousness over 10 minutes, scalp pathology, subject included in another clinical and/or therapeutic experiment in progress involving the testing of a therapeutic treatment or a drug treatment, opposition to participation in research, inability to perform cognitive tests: non-psychiatric (somatic) condition likely to affect cognitive abilities, sensory or peripheral motor deficits, clinical condition in acute phase (agitation, altered consciousness), protection of property measure such as safeguard of justice, healthy volunteers only: past or current severe psychiatric disorder (psychotic disorder, mood disorder (depressive and bipolar disorders), anxiety disorder, autism spectrum disorder and eating disorder).
* Sample: 360 subjects: 180 patients (30 subjects per group: (6 groups of 30 patients corresponding to severe psychiatric disorders: psychotic disorders, depressive disorders, bipolar disorders, anxiety disorders, autism spectrum disorders, eating disorders) and 180 healthy volunteers
* Procedure: After the patient / healthy volunteer has been informed about the study and has not objected to participating during a routine consultation, the patient / healthy volunteer will be included in the study. Cognitive tests will be collected as part of the patient's usual follow-up according to the pathology.
* Statistics: The different variables corresponding to the judgment criteria will be compared between the groups by being included as dependent variables in mixed linear regression models (ANOVA; or KRUSKAL-WALLIS if non-parametric) with the group as independent factor, time (before, after treatment) and type of treatment.
* Deliverables: constitution of a transnosographic atlas of neuro-cognitive deficits in different psychiatric pathologies.

ELIGIBILITY:
Inclusion criteria for patients:

* 18 to 65 years of age,
* Suffering from a severe psychiatric disorder (psychotic disorder, mood disorder (depressive and bipolar disorders), anxiety disorder, autism spectrum disorder and eating disorder),
* Benefiting from cognitive phenotyping (neuropsychological assessment and possibly EEG) as part of the initial assessment for a severe psychiatric disorder, proven non-opposition to participation in the study, ability to perform cognitive tests: speaking and understanding French easily, presence of an identified support person, absence or presence of a property protection measure such as curatorship or guardianship

Inclusion criteria for healthy volunteers:

* ages 18 to 65,
* proven non-opposition to participating in the study,
* ability to perform cognitive tests: able to speak and understand French

Exclusion criteria:

* impossible to collect information on exposure (subjects recently arrived in France, foreign language ...),
* history of coma, epilepsy, head trauma with loss of consciousness over 10 minutes, scalp pathology,
* subject included in another clinical and/or therapeutic experiment in progress involving the testing of a therapeutic treatment or a drug treatment,
* opposition to participation in research,
* inability to perform cognitive tests: non-psychiatric (somatic) condition likely to affect cognitive abilities, sensory or peripheral motor deficits, clinical condition in acute phase (agitation, altered consciousness),
* protection of property measure such as safeguard of justice,
* For healthy volunteers only: past or current severe psychiatric disorder (psychotic disorder, mood disorder (depressive and bipolar disorders), anxiety disorder, autism spectrum disorder and eating disorder).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Population : Patients with Severe Psychiatric Disorders (psychotic disorder, mood disorder (depressive and bipolar disorders), anxiety disorder, autism spectrum disorder and eating disorder) Control Population : Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
Main outcome | At inclusion
  The primary outcome is the comparison of cognitive-behavioral performance composite scores corresponding to response rates (in %) for each cognitive dimension between the different severe psychiatric disorder groups and the healthy subjects.

SECONDARY OUTCOMES:
Secondary outcome 1 | At inclusion
  Outcome will be the comparison of neurophysiological data from EEG recordings (composite variable) recorded simultaneously with the performance of behavioral tasks for each cognitive dimension between the different severe psychiatric disorders.
Secondary outcome 2 | Through study completion, up to 6 months
  Outcome will be the comparison of cognitive-behavioral performance composite score corresponding to response rates (in %) from neuropsychological tests before and after treatment (up to + 6 months) in the different groups of patients with severe psychiatric disorders.
Secondary outcome 3 | Through study completion, up to 6 months
  Outcome will be the comparison of neurophysiological data obtained from EEG recordings (composite variable) associated with behavioral tests before and after treatment (up to + 6 months) in the different groups of patients with severe psychiatric disorder.

IPD SHARING:
Plan to Share IPD: Undecided
Undecided